CLINICAL TRIAL: NCT03231384
Title: Safety and Feasibility of Rt-PA Thrombolytic Therapy in Combination With Remote Ischemic Conditioning for Acute Ischemic Stroke(rtPA-RIC1)
Brief Title: Rt-PA Thrombolytic Therapy in Combination With Remote Ischemic Conditioning for Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming, professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIC/rtPA
Record Dates: First submitted 2017-07-05; First posted 2017-07-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): The upper limb ischemic conditioning is composed of five cycles of upper limb ischemia intervened by reperfusion, which is induced by two cuff placed around the upper arms respectively and inflated to 200 mm Hg for 5 minutes followed by 5 minutes of reperfusion by cuff deflation. This therapy started within 2 hours after r-tPA thrombolytic therapy. In addition, all participants receive a standard clinical therapy.
  Interventions: Device: Remote ischemic conditioning
- Control group (No Intervention): The participants received r-tPA thrombolytic therapy after diagnosed ischemic stroke. In addition, all participants receive a standard clinical therapy.

INTERVENTIONS:
Device: Remote ischemic conditioning — In this study, the remote ischemic conditioning treatment was composed of five cycles of bilateral upper limb ischemia intervened by reperfusion, which was induced by two cuff placed around the upper arms respectively and inflated to 200 mm Hg for 5 minutes followed by 5 minutes of reperfusion by cuff deflation.
  Doctormate, IPC-906
  Arms: RIC group

SUMMARY:
The purpose of this study is to determine the safety and feasibility of remote limb ischemic conditioning(RIC) in acute ischemic stroke patients who received r-tPA thrombolytic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age≥18;
* Acute ischemic stroke;
* modified Rankin Scale (mRS) score of 2-5;
* mRS score less than 1 before onset of stroke symptom;
* Onset of stroke symptoms within 4.5h before initiation of intravenous rt-PA thrombolytic therapy;
* Good compliance for Remote Ischemic Conditioning(RIC) therapy;
* Informed consent obtained.

Exclusion Criteria:

* Stroke or serious head trauma within the previous 3 months
* Major surgery or severe trauma with in the preceding 3 months
* Intracranial hemorrhage
* Systolic pressure greater than 185 mm Hg or diastolic pressure greater than 110 mm Hg, or aggressive treatment intravenous medication) necessary to reduce blood pressure to these limits
* Symptoms rapidly improving
* Symptoms suggestive of subarachnoid hemorrhage, even if CT scan was normal
* Gastrointestinal hemorrhage or urinary tract hemorrhage within the previous 21 days
* Arterial puncture at a noncompressible site within the previous 7 days
* Seizure at the onset of stroke
* Platelet count of less than 100,000 per cubic millimeter
* Received heparin within the 48 hours preceding the onset of stroke and had an elevated partial-thromboplastin time
* Received oral anticoagulation therapy preceding the onset of stroke and INR greater than 1.7 or prothrombin times greater than 15 seconds
* CT showed a multiple infarction (low density area greater than 1/3 cerebral hemisphere)
* Use or plan to use intervention for diagnosis or treating
* Intracranial neoplasm, cerebral aneurysm or arteriovenous malformation
* severe hepatic or renal dysfunction
* Contraindication for remote ischemic conditioning: severe soft tissue injury, fracture, or peripheral vascular disease in the upper limbs.
* Life expectancy<1 years
* Pregnant or breast-feeding women
* Unwilling to be followed up or poor compliance for treatment
* Patients being enrolled or having been enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
Feasibility of RIC after acute ischemic stroke | 7 days
  The proportion of enrolled subjects that completed all the designed RIC procedures.

SECONDARY OUTCOMES:
Objective signs of tissue or neurovascular injury | within 7(±24h) days
  objective signs of tissue or neurovascular injury felt to be due to cuff inflation. Inspection included palpation of distal radial pulses, visual inspection (for local edema, redness, skin breakdown), and palpation for tenderness
Number of participants with intracranial hemorrhage in two groups | 7(±24h)days
Scores assessed by National Institutes of Health Stroke Scale(NIHSS) | 7(±24h)days
The functional outcome at 90 days assessed by modified Rankin scale (mRS). | 90( ±7days) days
functional outcome assessed by Barthel Index(BI) | 90( ±7days)days
cerebral infarct volume. | 3-7 days after stroke onset
  The infarct volume of cerebral infarct is evaluated by cranial noncontrast MRI
cerebral infarct volume. | 3-7 days after stroke onset
  The infarct volume of cerebral infarct is evaluated by cranial noncontrast CT
Cardiovascular parameters during 7 days of RIC treatment. | 7 days
  the blood pressure were measured immediately before RIC and also be measured 5 minutes after RIC.
the heart rate during 7 days of RIC treatment. | 7 days
  the heart rate were measured immediately before RIC and also be measured 5 minutes after RIC.
Levels of plasma myoglobin | baseline and 7(±2)days
Levels of serum IL-6 | baseline and 7(±2)days
Levels of serum HS-CRP | baseline and 7(±2)days
Levels of serum HCY | baseline and 7(±2)days
Any adverse events | 90(±7)days

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, XI Cheng District, China